CLINICAL TRIAL: NCT00353106
Title: The Experience of Having Chronic Graft-Versus-Host Disease
Brief Title: Experience of Having Chronic Graft-Versus-Host Disease
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2005-0727
Record Dates: First submitted 2006-07-13; First posted 2006-07-17 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Graft-Versus-Host Disease
Keywords: Graft-Versus-Host Disease; GVHD; Chronic Graft-Versus-Host Disease; cGVHD; Interview; Questionnaire; Survey; Caregiver
MeSH Terms: conditions — Graft vs Host Disease; Bronchiolitis Obliterans Syndrome | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients: Patients with chronic GVHD
  Interventions: Behavioral: Interview; Behavioral: Questionnaire
- Content Expert Panel: Content expert panel with 5 years experience caring for patients with cGVHD.
  Interventions: Behavioral: Questionnaire
- Caregivers: Caregivers of patients with cGVHD
  Interventions: Behavioral: Interview; Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Interview — 30-minute interviews of participating patients and their caregiver(s).
  Groups: Caregivers; Patients
Behavioral: Questionnaire — Questionnaires that will take approximately 5 minutes to complete.
  Other Names: Survey

SUMMARY:
Primary Objectives:

1. To explore the experience of chronic graft-versus-host disease (cGVHD) following allogeneic blood or marrow transplantation from the perspective of the patient and the patient's primary family caregiver.
2. To develop and validate an instrument to measure the severity of multiple symptoms and the impact of these symptoms on daily functioning in patients who have cGVHD.

Secondary Objectives:

1. To develop a detailed description of the experience of having cGVHD.
2. To develop a detailed description of the symptom experience of cGVHD to allow for development of a symptoms instrument for cGVHD.
3. To assess the understanding of questions to measure the symptoms of cGVHD in patients with various levels of education.
4. To develop a detailed description of caring for a patient with cGVHD.

DETAILED DESCRIPTION:
For Patient:

If you agree to take part in this study, you will be asked to take part in 1 interview. During the interview, you will be asked to describe what it has been like for you to have chronic GVHD. In addition, if you agree to take part in this study, your family caregiver, if you have one, will be approached to take part in the study.

For Caregiver:

If you agree to take part in this study, you will be asked to take part in 1 interview. During the interview, you will be asked to describe what it has been like for you to help care for a family member with chronic GVHD.

Both Parties:

The interview face-to-face will take place while you are at M. D. Anderson receiving care. You will be interviewed alone and the information gathered during the interview will be strictly confidential. The interview will take about 30 minutes and will be tape recorded. The audiotape of the interview will be kept in a locked cabinet in the office of the study chairperson Dr. Loretta Williams. If other study personnel need the tape for analysis, they must obtain the tape directly from Dr. Williams. They may keep the tape only while they are listening to it and must return it immediately to Dr. Williams. Identification labels on the tape will only contain your study number and will not contain your name, medical record number, or other identifying information. When all analysis for the study has been completed and reported, the audiotape will be destroyed.

After the interview, you will be asked to answer a face-to-face questionnaire. This questionnaire will ask descriptive personal information (age, marital status, etc.). Answering these questions should take about 5 minutes.

Your participation on this study ends after you complete the interview and questionnaire.

This is an investigational study. About 20 patients and 20 caregivers will take part in this study. All will be enrolled at M. D. Anderson.

For Patient - Phase III:

If you agree to take part in this study, you will be asked to complete 1 questionnaire. The questionnaire will have questions asking you to rate how severe your current symptoms are and how much these symptoms disrupt your daily activities. You will be asked to complete this questionnaire during your clinic visit. The questionnaire will take no more than 10 minutes to complete.

If you have chronic graft-versus-host disease, you will be asked to complete a second questionnaire about your opinion of the symptom questionnaire (the first questionnaire). For example, you will be asked if the symptom questionnaire was easy to understand and to complete. Learning your opinion about this questionnaire will help researchers learn what important questions may be missing from the questionnaire. The questionnaire will take no more than 10 minutes to complete.

If you have chronic graft-versus-host disease, you will also be given questions asking you to rate the overall quality of your life and your ability to function. These ratings should take no more than 2 minutes to complete.

Finally, you will be asked to answer a questionnaire. This questionnaire will ask descriptive personal information (such as age and marital status). Answering these questions should take about 5 minutes.

If you have chronic GVHD, you may be asked to fill out the questionnaire rating your symptoms 1 more time, about 3 days after you completed it the first time. You will return this second questionnaire to the research staff in a pre-addressed, stamped envelope given to you by the research staff. If you are asked to complete the questionnaire this second time, the research staff will also ask for your telephone number so that they may contact you and remind you to complete the questionnaire.

Identification labels on all study questionnaires and forms will only contain your study number and will not contain your name, medical record number, or other identifying information. All study materials will be kept in a locked cabinet at all times. When all analysis for the study has been completed and reported, the questionnaires will be destroyed.

The study ends when you have completed the questionnaires, rating scales, and interview in the clinic, or when you have completed and returned the second questionnaire 3 days after your clinic visit.

This is an investigational study. Up to 192 patients will take part in this study. 147 will be enrolled at M. D. Anderson and 45 will be enrolled at Roswell Park Cancer Institute.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Ability to speak and read English
3. Clinical or histological diagnosis of active cGVHD or at least 3 months post allogeneic BMT without a diagnosis of active GVHD (PATIENT ONLY)
4. Identification as the single primary family caregiver by a patient with cGVHD (CAREGIVER ONLY)
5. Physician or nurse with at least 5 years experience caring for patients with cGHVD (PROFESSIONAL EXPERT ONLY)
6. At least one publication in the last 5 years dealing with cGVHD (PHYSICIAN PROFESSIONAL EXPERT ONLY)
7. Consent to participate

Exclusion Criteria:

1. Inability to understand the intent of the study
2. Medical condition that would preclude participation in an interview lasting 30 minutes (PHASE 1 OF STUDY ONLY)
3. Diagnosis of active psychosis or severe cognitive impairment
4. Bone marrow or stem cell donor for patient (CAREGIVER ONLY)
5. Disease for which BMT was performed not in remission (PATIENT ONLY)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants with chronic graft-versus-host disease (cGVHD) following allogeneic blood or marrow transplantation, the patient's primary family caregiver, and content expert panel.
Sampling Method: Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2006-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Phase 1: Open-Ended Interview/Questions designed to elicit specific descriptions of experience of having cGVHD or caring for a patient with cGVHD | At time of treatment, duration approximately 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Loretta A. Williams, DSN, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - UT MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org